CLINICAL TRIAL: NCT03283878
Title: Perioperative Antibiotic Prophylaxis in Patients Undergoing Elective Total Knee Arthroplasty: A Prospective, Randomized, Open-label, Controlled Multi-center Trial
Brief Title: Antibiotic Prophylaxis in Patients Undergoing Elective Total Knee Arthroplasty- Multi-center Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Association of Hip and Knee Surgeons (Other); Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00086892
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arthropathy of Knee; Antibiotic Prophylaxis
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group 1 (Experimental): Patients in Group #1 will receive a single weight-based dose of prophylactic cefazolin antibiotic that is administered intravenously within less than 60 minutes prior to skin incision in elective total knee arthroplasty. No further antibiotic administration will be given.
  < 120 kg - patients will receive 2 grams of cefazolin
  ≥ 120 kg - patient will receive 3 grams of cefazolin
  Patients with documented allergy/anaphylactic reaction to penicillin or cephalosporin may receive intravenous vancomycin monotherapy or dual therapy with vancomycin and gentamicin as an alternative. In addition, the use of clindamycin as an alternative is also permitted at a minimum recommended dose.
  Interventions: Drug: Cefazolin
- Study Group 2 (Experimental): Patients in Group #2 will receive a single weight-based dose of prophylactic cefazolin antibiotic that is administered intravenously within less than 60 minutes prior to skin incision in elective total knee arthroplasty. In addition, two weight-based doses of cefazolin will be administered within 24 hours postoperatively.
  < 120 kg - patients will receive 2 grams of cefazolin
  ≥ 120 kg - patient will receive 3 grams of cefazolin
  Patients with documented allergy/anaphylactic reaction to penicillin or cephalosporin may receive intravenous vancomycin monotherapy or dual therapy with vancomycin and gentamicin as an alternative. If allergic, patients will also receive two weight-based doses vancomycin postoperatively but not gentamicin postoperatively. In addition, the use of clindamycin as an alternative is also permitted. Vancomycin schedule: one dose preoperatively, one dose 8-12 h postoperatively, one dose 24 h postoperatively (opt.).
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin will be administered intravenously within less than 60 minutes prior to skin incision in elective TKA for Group 1.
  Cefazolin will be administered intravenously within less than 60 minutes prior to skin incision in elective TKA. In addition, two weight based doses of cefazolin will be administered within 24 hours postoperatively for Group 2.
  Other Names: Ancef

SUMMARY:
The Antibiotic Prophylaxis in Patients Undergoing Elective Total Knee Arthroplasty (TKA): Multi-Center Trial is a study that will compare the effectiveness of various perioperative strategies for antibiotic delivery as prophylaxis for periprosthetic joint infections (PJI) and surgical site infection in elective primary TKA. The investigators hypothesize that a single dose of prophylactic antibiotic administered within 60 minutes before the incision is not an effective way to prevent PJI in elective primary total knee arthroplasty (TKA). The investigators also hypothesize that the prolonged delivery (24 hours) of antibiotic prophylaxis after surgery does not further reduce the incidence of PJI in elective primary TKA.

Duke University is the only site recruiting both primary total knee arthroplasty and unilateral knee arthroplasty.

DETAILED DESCRIPTION:
Total joint arthroplasty (TJA), is one of the most successful operations in modern medicine; however, it remains an expensive procedure in an era of constrained health care resources. Arthritis affects 49.9 million Americans with 21.1 million experiencing arthritis-attributable activity limitations. As these numbers are expected to increase significantly by 2030, the demand for primary total knee arthroplasties (TKA) by 673% to 3.48 million procedures/year. Periprosthetic joint infection (PJI), with its disastrous implications, continues to challenge the orthopaedic community. Practicing orthopaedic surgeons continue to invest efforts to minimize surgical site infection (SSI). Kamath et al. evaluated characteristics and resource utilization associated with revision arthroplasty for PJI using the Nationwide Inpatient Sample. The authors found that PJI was the most common indication for revision total knee arthroplasty (TKA), and the third most common reason for revision total hip arthroplasty (THA). Prophylactic antibiotics aim to provide protection against bacteria most likely to gain access to the surgical site during the procedure and in the perioperative period. The two most common bacteria causing contamination and subsequent deep infection in TKA are Staphylococcus aureus and coagulase-negative staphylococci.

While antibiotic regimens for antimicrobial prophylaxis might carry different risks and side-effect profiles, e.g., hypersensitivity reactions (including anaphylaxis), acute kidney injury, and Clostridium difficile infection, there are a number of studies which validate the importance of the preoperative dose of antibiotics in decreasing periprosthetic joint infection (PJI) and surgical site infection (SSI) in total joint arthroplasty (TJA). However, there are conflicting recommendations/guidelines as to the optimal timing and the optimal duration perioperative antibiotics. The American Academy of Orthopaedic Surgeons (AAOS), the Centers for Disease Control (CDC), and SCIP guidelines recommend that prophylactic antibiotics be completely infused within one hour before the surgical incision. The US advisory statement recommends that antimicrobial prophylaxis be administered within one hour before incision and discontinued within 24 hours after the end of the operation, while European guidelines recommend a single dose within 30 minutes before incision.

Recently, the Center for Disease Control (CDC) published its updated guidelines for prevention of SSI prevention that included a recommendation regarding peri-operative antibiotic prophylaxis. Based on their evaluation of the available literature, the CDC recommended that a single dose of peri-operative antibiotics be utilized for patients undergoing clean-contaminated surgical interventions, advocating for no prophylaxis after the incision is closed in the operating room. This guideline encompasses several surgeries where implants are utilized, including arthroplasty, spine fusion, and fracture fixation. Furthermore, it was classified as a category IA-strong recommendation with high quality evidence. However, much of the literature cited for this recommendation is based on cardiothoracic, vascular, and general surgeries, where few or no implants are utilized. It is important to recognize that these surgical cohort may behave differently from the orthopaedic patient population in terms of infection risk and severity of infection outcomes.

This clinical research protocol seeks to address the lack of knowledge and Level I data around the optimal antimicrobial prophylaxis and to address the question if a single preoperative dose is enough compared to additional postoperative prophylaxis. Several smaller clinical studies have used pre- and post-intervention periods to assess the effect of antibiotic duration for surgical prophylaxis. Tang et al launched a surgical wound infection surveillance program to monitor all orthopaedic surgeries and changed the prophylactic antibiotic regimen from intravenous cefuroxime (one preoperative and 2 postoperative doses every 8 hours) to one single preoperative dose of intravenous cefazolin for all clean orthopaedic surgeries. The authors of this study found no significant difference in the superficial and deep wound infection rates in 1,367 primary arthroplasties performed with a single preoperative dose of cefazolin versus 3 doses of cefuroxime. The deep wound infection rate for THA was 1.1% (95% CI, 0%-3.3%) in the cefuroxime group and 1.1% (95% CI, 0%-2.2%) in the cefazolin group (p=1.0). The deep wound infection rate of TKA was 1.6% (95% CI, 0%-3.8%) in the cefuroxime group and 1.0% (95% CI, 0.3%-1.7%) in the cefazolin group (p=0.63).121 In a retrospective review of 1,341 TJAs, Williams and Gustilo found no difference in deep infection rates between a 3 day and 1 day course of prophylactic antibiotics, but emphasized the importance of the preoperative dose, which was 2g of cefazolin. Mauerhan compared the efficacy of a one-day regimen of cefuroxime with a 3-day regimen of cefazolin in a prospective, double-blinded, multicenter study of 1,354 patients treated with arthroplasty and concluded that there was no significant difference in the prevalence of wound infections between the two groups.[34] In the group treated with primary THA, the prevalence of deep wound infection was 0.5% (1/187) for those treated with cefuroxime compared with 1.2% (2/168) for those who had received cefazolin. In the group treated with a primary TKA, the rate of deep wound infection was 0.6% (1/178) for those treated with cefuroxime compared with 1.4% (3/207) for those who had received cefazolin. Heydemann and Nelson, in a study of hip and knee arthroplasty procedures, initially compared a 24-hour regimen of either nafcillin or cefazolin with a 7-day regimen of the same and found no difference in the prevalence of infection. They then compared a single preoperative dose with a 48-hour regimen and again found no difference in infection prevalence. A total of 466 procedures was performed during the 4-year study. No deep infections developed in either the one-dose or 48-hour antibiotic protocol group. A deep infection developed in one (0.8%) of the 127 patients in the 24-hour protocol group and in two (1.6%) of the 128 patients in the 7-day protocol group for an overall infection rate of 0.6% (3/466). The authors recognized that as a result of the small sample sizes, the study lacked the power to compare the one dose and the more than one dose categories. In two trials, a total of 1609 patients were randomly assigned to receive 1.5 g of cefuroxime intravenously every 8 hours for a total of 16 hours (n = 1511) or 24 hours (n = 98) postoperatively versus 1600 patients given no postoperative prophylaxis. Both studies showed no difference between treatment groups suggesting that current available evidence may not support the efficacy of postoperative antibiotic prophylaxis for the prevention of surgical-site infections.

Antibiotics have been a critical public health tool since the discovery of penicillin in 1928, saving the lives of millions of people around the world. Today, however, the emergence of drug resistance in bacteria is reversing the miracles of the past eighty years, with drug choices for the treatment of many bacterial infections becoming increasingly limited, expensive, and, in some cases, nonexistent. The Centers for Disease Control and Prevention (CDC) estimates that drug-resistant bacteria cause two million illnesses and approximately 23,000 deaths each year in the United States alone. The Centers for Disease Control and Prevention (CDC) estimates that drug-resistant bacteria cause two million illnesses and approximately 23,000 deaths each year in the United States alone (https://www.cdc.gov/drugresistance/). The National Action Plan for Combating Antibiotic-resistant Bacteria provides a roadmap to guide the Nation in rising to this challenge. Developed in response to Executive Order 13676: Combating Antibiotic-Resistant Bacteria - issued by President Barack Obama on September 18, 2014 - the National Action Plan outlines steps for implementing the National Strategy for Combating Antibiotic-Resistant Bacteria and addressing the policy recommendations with regard to antibiotic stewardship as outlined by the President's Council of Advisors on Science and Technology (PCAST). One of the goals of the National Action Plan is the implementation of evidence-based infection control practices can prevent the spread of resistant pathogens and questions the way surgeons use prophylactic antibiotics in the preoperative period.

The scientific rationale for antibiotic prophylaxis is to inhibit or eliminate contaminating microorganisms that gain access to the surgical site during the procedure. Thus, the goal of administering preoperative antibiotics is to allow for adequate tissue (blood, soft tissue, and bone) concentrations by the time of incision. Thus, these antibiotics should exceed the minimum inhibitory concentration (MIC) for the organisms most likely to be encountered for the duration of the operation. While the role of perioperative antibiotic prophylaxis is well established, controversy exists about best clinical practice guidelines with regard to antibiotic regimen and route of administration. The results of the proposed study will be used to establish a clinical practice guidelines for antimicrobial prophylaxis in elective total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age
* Patient has no open wounds on operative leg
* Patient is scheduled to undergo elective total knee arthroplasty for posttraumatic, osteoarthritis, avascular necrosis, and/or inflammatory arthritis
* Patient does not have active infection on the operative leg, the operative joint
* Patient is willing to cooperate and follow study protocol and visit schedule

Exclusion Criteria:

* Patient is ≤ 18 years of age
* Patient is pregnant
* Patient is unable to provide written consent
* Patient has psychiatric disorder that precludes safe study participation or that necessitates confinement in a custodial environment at home or in a chronic care facility
* Patient has traumatic injury that requires emergent or urgent total knee arthroplasty (e.g. fracture)
* Patient has active infections in the operative leg/joint
* Patient has severe dementia
* Suspicion of illicit drug abuse by patient. Patients who use prescription cannabinoids are not excluded from enrollment.
* ASA score of 5 & 6
* No application of topical antibiotic powder such as vancomycin or antibiotic beads in surgical wound
* Intra-operative re-dosing other than specified re-dosing intervals or without excessive blood loss (<1500mL)
* History of prior native septic knee arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1770 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Rate of periprosthetic infection (PJI) as measured by chart review | 90 day post-op

SECONDARY OUTCOMES:
Costs of antibiotic treatment as measured by costs summed over all patients and divided by group size | up to 1 year

OTHER OUTCOMES:
Rate of periprosthetic infection (PJI) as measured by phone call, email, letter and/or secured messaging via electronical medical record system | 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Seyler, MD, Principal Investigator — Duke University
Locations (14):
- United States (14):
  - University of California, San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - University of Maryland St. Joseph Medical Center & Orthopedic Associates, Towson, Maryland
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Mississippi Bone and Joint Clinic, Starkville, Mississippi
  - University Orthopaedic Associates, LLC, Somerset, New Jersey
  - NYU School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - BaylorScott&White Research Institute, Temple, Texas
  - Augusta Health, Fishersville, Virginia